CLINICAL TRIAL: NCT04865861
Title: The Characteristic of Airway Microbiome Profiling of Chronic Obstructive Pulmonary Disease-bronchiectasis Overlap Patients and Its Association With Acute Exacerbation
Brief Title: The Characteristic of Airway Microbiome Profiling of COPD-bronchiectasis Overlap Patients and Its Association With Acute Exacerbation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Zhenfeng He, Principle investigator, Guangzhou Medical University
Other Study IDs: GIRH-2020-156
Record Dates: First submitted 2021-04-25; First posted 2021-04-29 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Bronchiectasis Adult; Chronic Obstructive Pulmonary Disease; Overlap; Microbiome
Keywords: Bronchiectasis; Chronic Obstructive Pulmonary Disease; overlap; microbiome; exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchiectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — serum; plasma; blood cell; sputum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overlap between chronic obstructive pulmonary disease (COPD) and bronchiectasis is a neglected area of research, and it is not covered by guidelines for clinical practice.

COPD and bronchiectasis share common symptoms of cough with sputum production and susceptibility to recurrent exacerbations driven by new or persistent infection.

Physiological criteria for the diagnosis of COPD and structural criteria for the diagnosis of bronchiectasis create the possibility for individual patients to fulfil both, resulting conceptually in either co-diagnosis or an overlap syndrome between the two conditions. The prevalence of this overlap will vary depending on the respective prevalence of COPD and bronchiectasis in the population under consideration.

A recent study of 201 COPD patients with airway wall abnormalities typical of bronchiectasis confirmed an association with exacerbations and was predictive of mortality over 48 months. A further, single-centre study demonstrated a near three-fold increased mortality rate, with patients with bronchiectasis and associated COPD having a 5-year mortality of 55%, compared with 20% in those with bronchiectasis without COPD. Airflow obstruction is perhaps best considered one marker of disease severity in bronchiectasis.

Disease-associated exacerbations have a major effect on patient healthcare costs as well as quality of life due to increased lung damage and mortality risk. Microorganisms such as Pseudomonas aeruginosa and, to a lesser extent, other Gram-negative and Gram-positive microorganisms identified in culture, have been linked to disease progression, poor clinical outcomes in bronchiectasis and driving airway neutrophil-mediated inflammation. The microbiome has the potential to provide valuable information regarding disease phenotype/endotype, treatment responses and targets for future therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as COPD, bronchiectasis or overlap based on HRCT and lung function test.
* Aged between 18 and 80 years.

Exclusion Criteria:

* Patients with active tuberculosis, traction bronchiectasis, malignancy, and severe systemic diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a single-center prospective observational study in which we will enroll the patients diagnosed as COPD, bronchiectasis or overlap (with or without chronic cough, daily sputum production) from the First Affiliated Hospital of Guangzhou Medical University between May 2020 and June 2023.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
The number of exacerbation events | 1 year
  The exacerbation of bronchiectasis is defined as a deterioration in three or more of the following key symptoms for at least 48 h: cough; sputum volume and/or consistency; sputum purulence; breathlessness and/or exercise tolerance; fatigue and/or malaise; haemoptysis AND a clinician determines that a change in bronchiectasis treatment is required.

SECONDARY OUTCOMES:
α-diversity | 1 hour
  α-diversity is a measure of how diverse a sample is based on how many species here are (richness) and how abundant each species is (evenness) within that sample.
β-diversity | 1 hour
  β-diversity is used to show how different samples are from each other, based on ifferences in bacterial presence, abundance or a phylogenetic tree
The positive result of bacteria culture and viral PCR. | 1 hour
  The positive result of bacteria is defined as at least one positive potentially-pathogenic bacteria being cultured from sputum (Haemophilus influenzae, Moraxella catarrhalis, Streptococcus pneumoniae, Pseudomonas aeruginosa, or Staphylococcus aureus).
  The positive result of viral is defined as at least one positive viral PCR (HRV, RSV, influenza virus, parainfluenza virus, human metapneumovirus, adenovirus, human bocavirus, or coronavirus) from sputum.

CONTACTS AND LOCATIONS:
Overall Officials: Weijie Guan, PhD, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University; Nanshan Zhong, PhD, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University., Guangzhou, Guangdong, China